CLINICAL TRIAL: NCT04713397
Title: Leg Length Discrepancy and Adolescent Idiopathic Scoliosis: Clinical and Radiological Characteristics
Status: Completed | Type: Observational
Sponsor: Hürriyet Yılmaz (Other)
Collaborators: Medipol University (Other); Dokuz Eylul University (Other); Başakşehir Çam & Sakura City Hospital (Other Government)
Responsible Party: Sponsor-Investigator, Hürriyet Yılmaz, MD.Prof., Halic University
Organization: Halic University (Other)
Other Study IDs: HUEK171-30
Record Dates: First submitted 2021-01-14; First posted 2021-01-19 (Actual); Last update posted 2021-05-24 (Actual); Status verified 2021-01

CONDITIONS: Leg Length Inequality; Scoliosis; Pelvic Obliquity
Keywords: Leg Length Discrepancy; Adolescent Idiopathic Scoliosis; Leg Length Discrepancy Scoliometer Test
MeSH Terms: conditions — Leg Length Inequality; Scoliosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- LLD group: Patients who have functional scoliosis due to structural LLD
  Interventions: Diagnostic Test: Leg Length Discrepancy Scoliometer Test
- LLD concurrent with AIS: Patients who have structural LLD concurrent with AIS
  Interventions: Diagnostic Test: Leg Length Discrepancy Scoliometer Test

INTERVENTIONS:
Diagnostic Test: Leg Length Discrepancy Scoliometer Test — A scoliometer used as an indirect and quantitative method to evaluate LLD for the first time in this study, and described it as "Leg Length Discrepancy Scoliometer Test". Scoliometer were used on Adams' forward bending position and the level of the pelvis accepted as equal when the scoliometer degree pointed zero on the sacral basis (angle of trunk rotation on sacrum). When considering pelvis level is high on the longer side and is low on the shorter side, if the angle of the scoliometer on the sacrum is negative (slope to the left), the left extremity was considered as shorter. In order to determine its correlation with an indirect method, scoliometer degree on the sacral basis was recorded then wooden blocks were added to the unequal leg side on the sacral basis until the pelvic equality was achieved on the scoliometer. Afterward, a correlation between the first measurement of ATRsacrum and the height of the wooden block which provides ATRsacrum to reach zero was investigated.

SUMMARY:
The aim of this retrospective study is to present clinical and radiological features and their relationships for differentiating functional scoliosis due to LLD and LLD concurrent with AIS.

DETAILED DESCRIPTION:
This study was conducted as a single-center retrospective comparative study on 47 consecutive scoliosis patients detected LLD, aged 10-18 years, between 2018 and 2020. The scoliosis patients with a diagnosis of structural LLD were divided into two groups according to whether there was a concurrent AIS diagnosis or not. Demographic data were recorded. Limb length was clinically measured by direct, indirect evaluation method and new LLD-Scoliometer Test. Cobb degree, axial rotation, internal/external pelvic obliquity and LLD were obtained from posteroanterior spine radiographs measured by two blinded orthopaedic spine surgeons.

ELIGIBILITY:
Inclusion Criteria:

* Between December 2018-2020
* Scoliotic patients, who detected LLD
* Ages 10 to 18 years
* Patients who have two or more clinical records at least 6 months apart
* Who accepted to participate in the study.

Exclusion Criteria:

* Neurological disease
* A history of spinal surgery/tumors
* The diagnosis of AIS without LLD or trauma

Ages: 10 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: 10 to 18 years scoliotic patients diagnosed with structural LLD
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2019-01-06 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2021-01-30 (Actual)

PRIMARY OUTCOMES:
Full spine PA radiography | baseline
  Posteroanterior whole spine digital X-Ray images were obtained with the patient barefoot, both heels on the floor, and both knees extended in an upright standing position. The digital radiography detector was 350x430 millimeters in size and clearly showed the positions of the femoral heads, the iliac crests, and whole spine. The distance between the X-ray tube and the detector was two meters. All radiographic data such as Cobb degree, axial rotation by Perdriolle and pelvic obliquity were measured by two blinded orthopaedic spine surgeons using Surgimap ® Spine (Nemaris ™ Inc, New York, NY) a validated software
direct evaluation- tape measure | baseline
  Limb length was clinically with a tape measure while the patient was in a supine position. For the direct evaluation method, measurements were taken from the anterior superior iliac spine to the medial malleolus.
indirect evaluation- wooden blocks | baseline
  indirect evaluation method, wooden blocks of known height were used to evaluate the amount of LLD in standing position.

CONTACTS AND LOCATIONS:
Overall Officials: Ahsen Büyükaslan, PT, PhD(c), Principal Investigator — Medipol University; Kadir Abul, MD, Study Chair — Başakşehir Çam & Sakura City Hospital; Haluk Berk, MD, Prof., Study Director — Dokuz Eylul University; Hürriyet Yilmaz, MD, Prof., Study Director — Halic University
Locations (1):
- Formed Healthcare Scoliosis Treatment and Brace Center, Istanbul, Sisli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Buyukaslan A, Abul K, Berk H, Yilmaz H. Leg length discrepancy and adolescent idiopathic scoliosis: clinical and radiological characteristics. Spine Deform. 2022 Mar;10(2):307-314. doi: 10.1007/s43390-021-00417-0. Epub 2021 Sep 28. PMID 34581993